CLINICAL TRIAL: NCT02307344
Title: Effect of Nigella Sativa on Nonalcoholic Steatohepatitis and Steatosis
Acronym: NASH NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0002-14-HYMC
Record Dates: First submitted 2014-11-03; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Nonalcoholic Steatohepatitis; Liver Steatosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nigella Sativa Supplement (Active Comparator): Fifty patients suffering from Nonalcoholic Steatohepatitis or Liver Steatosis will ingest capsules containing 2 grams of Nigella Sativa divided into 1 grams twice a day.
  Interventions: Dietary Supplement: Nigella Sativa
- Patients receiving a placebo tablet (Active Comparator): Twenty patients suffering from Nonalcoholic Steatohepatitis or Liver Steatosis will ingest placebo capsules twice a day, that look like the capsules of those receiving the Nigella Sativa.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nigella Sativa
  Arms: Nigella Sativa Supplement
Dietary Supplement: Placebo — Capsules that contain a placebo but look like the Nigella Sativa capsules
  Arms: Patients receiving a placebo tablet

SUMMARY:
The investigators hypothesize that Nigella Sativa will have an effect on Nonalcoholic Steatohepatitis and Liver Steatosis by enhancing lipophagy in the liver tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Steatohepatitis
* Patients suffering from Liver Steatosis

Exclusion Criteria:

* Patients suffering from viral hepatitis
* Patients with HIV infection
* Patients suffering from Wilsons Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Nigella Sativa on Liver Triglyceride Concentration | One year
  The difference in change in the average liver triglyceride concentration will be measured by MRI Spectroscopy between the Nigella Sativa arm and the placebo arm, at start and end of the study.

SECONDARY OUTCOMES:
Effect of Nigella Sativa on Improvement in NASH Activity Index | One year
  Improvement in Nash activity Index will be measured by the NAFLD Activity Score.
Effect of Nigella Sativa on Fibrosis Staging | One year
  Microscopic examination of two liver biopsies at start and end of the study, to determine fibrosis staging.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel